CLINICAL TRIAL: NCT02044393
Title: Relative Bioavailability of a Single Oral Dose of BI 691751 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, Randomised, Two-period, Two-sequence Crossover Study)
Brief Title: Interaction of BI 691751 With Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1334.10; 2013-003814-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

ARMS (2):
- Reference (Experimental): single dose BI 691751
  Interventions: Drug: BI 691751
- Test (Experimental): multiple doses of itraconazole + single dose BI 691751
  Interventions: Drug: itraconazole; Drug: BI 691751

INTERVENTIONS:
Drug: itraconazole — multiple doses of itraconazole given as capsules
  Arms: Test
Drug: BI 691751 — single dose BI 691751 given as tablet
  Arms: Test
Drug: BI 691751 — single dose BI 691751 given as tablet
  Arms: Reference

SUMMARY:
Investigation of the relative bioavailability of a single dose of BI 691751 when given alone and together with itraconazole; safety and tolerability

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. body mass index (BMI) of 18.5 to 29.9 kg/m2
3. Subjects must be able to understand and comply with study requirements

Exclusion criteria:

1. Any finding in the medical examination (including blood pressure (BP), pulse rate (PR), or electrocardiogram (ECG)) deviating from normal and judged clinically relevant by the investigator.
2. Pulse rate outside 45 to 100 bpm or repeated measurements of systolic BP outside 90 to 140 mmHg or diastolic BP outside 50 to 90 mmHg.
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any alanine transaminase (ALT/GPT), aspartate transaminase (AST/GOT), or gammaglutamyltransferase (GGT) value outside the reference range at the screening examination
5. Any evidence of a concomitant disease judged clinically relevant by the investigator
6. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
7. Any history of relevant liver diseases such as disturbance of liver function, jaundice, drug induced liver injury, Dubin-Johnson syndrome, Rotor syndrome, or liver tumors

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1334.10.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole (IT) +BI 691751 / BI 691751: Subjects in treatment sequence of tested drug treatment in period 1, then reference drug treatment in period 2 (T/R): two capsules of 100 mg itraconazole were given twice daily on Day -3 (loading dose) and once daily on Day -2 to Day 7 (10 days of itraconazol treatment in total). In addition, 1 tablet of 10 mg BI 691751 was given as a single dose on Day 1 (corresponding to the fourth day of the 10-day itraconazole treatment) in period 1. One tablet of 10 mg BI 691751 was given as a single dose on Day 1 in period 2.
  The BI 691751 single dose administrations in the 2 treatment periods were separated by a washout period of at least 7 weeks.
  Oral administration with 240 mL water after intake of a standardised meal.
- BI 691751 / IT+BI 691751: Subjects in treatment sequence of reference drug treatment in period 1, then tested drug treatment in period 2 (R/T): One tablet of 10 mg BI 691751 was given as a single dose on Day 1 in period 1. Two capsules of 100 mg itraconazole were given twice daily on Day -3 (loading dose) and once daily on Day -2 to Day 7 (10 days of itraconazol treatment in total), and, 1 tablet of 10 mg BI 691751 was given as a single dose on Day 1 (corresponding to the fourth day of the 10-day itraconazole treatment) in period 2.
  Oral administration with 240 mL water after intake of a standaridsed meal.
Period: Period 1
Arm/Group | Itraconazole (IT) +BI 691751 / BI 691751 | BI 691751 / IT+BI 691751
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Itraconazole (IT) +BI 691751 / BI 691751 | BI 691751 / IT+BI 691751
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): included all subjects who were randomized and took at least one dose of study medication during the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Itraconazole (IT) +BI 691751 / BI 691751 | BI 691751 / IT+BI 691751 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.9) | 37.4 (6.6) | 36.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of BI 691751 in Plasma and Whole Blood Over the Time Interval From 0 up to the Last Quantifiable Concentration)
Description: AUC0-tz: area under the concentration-time curve of BI 691751 in plasma and whole blood over the time interval from 0 up to the last quantifiable concentration.
Time Frame: from day 1 to 31 days postdose relative to BI 691751 administration (h:min): -2:00, 0:10, 0:20, 0:40, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00, 34:00, 47:00, 71:00, 95:00, 119:00, 143:00, 215:00, 287:00, 383:00, 551:00, 719:00h.
Population: Pharmacokinetic Set (PKS): included all subjects from the TS who provided at least one primary or secondary pharmacokinetic endpoint in any period that is judged as evaluable for pharmacokinetics and is not affected by protocol violations relevant to the statistical evaluation of bioavailability
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- BI 691751: single dose BI 691751
  BI 691751: 10 mg single dose oral administration with 240 mL water after intake of a standard meal.
- IT + BI 691751: Two capsules of 100 mg IT were given twice daily on Day -3 and once daily on Day -2 to Day 7. 1 tablet of 10 mg BI 691751 was given as a single dose on Day 1 with 240 mL water after intake of a standard meal.
Arm/Group | BI 691751 | IT + BI 691751
Number analyzed (Participants) | 20 | 20
nmol*h/L
  in plasma | 2830 (34.6) | 2090 (43.2)
  in whole blood | 25000 (25.8) | 21600 (25.8)
Statistical Analysis 1: Comparison: BI 691751 vs IT + BI 691751; gMean ratio of IT+BI 691751 to BI 69175 treatment (in plasma); Test type: Non-Inferiority or Equivalence — 90% confidence interval for gMean ratio of IT+BI 691751 to BI 69175 treatment was provided. The ANOVA model included the fixed effects 'sequence', 'period' and 'treatment' and as a random effect 'subject within sequence' as source of variation; gMean ratio = 74.07, 90% CI 2-sided [62.371 to 87.959], Standard Error of Mean 32.1 — ratio of IT+BI 691751 to BI 691751 treatment. Estimated value and its confidence interval (CI) are in percentage unit. The standard error of the mean actually is the geometric coefficient of variance
Statistical Analysis 2: Comparison: BI 691751 vs IT + BI 691751; gMean ratio of IT+BI 691751 to BI 691751 treatment (in whole blood); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean ratio = 86.35, 90% CI 2-sided [78.04 to 95.56], Standard Error of Mean 18.6 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Cmax (Maximum Measured Concentration of BI 691751 in Plasma and Whole Blood)
Description: Cmax (maximum measured concentration of BI 691751 in plasma and whole blood).
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- BI 691751: 10 mg BI 691751 single dose oral administration with 240 mL water after intake of a standard meal.
Arm/Group | BI 691751 | IT + BI 691751
Number analyzed (Participants) | 20 | 20
nmol/L
  in plasma | 157 (24.4) | 150 (34.1)
  in whole blood | 217 (16.0) | 203 (21.4)
Statistical Analysis 1: Comparison: BI 691751 vs IT + BI 691751; gMean ratio of test to reference treatment (in plasma); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean ratio = 95.59, 90% CI 2-sided [84.195 to 108.537], Standard Error of Mean 23.5 — ratio of test to reference treatment. The standard error of the mean actually is the geometric coefficient of variance
Statistical Analysis 2: Comparison: BI 691751 vs IT + BI 691751; gMean ratio of test to reference treatment (in whole blood); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean ratio = 93.54, 90% CI 2-sided [86.142 to 101.570], Standard Error of Mean 15.1 — ratio of test to reference treatment. The standard error of the mean actually is the geometric coefficient of variance

3. Secondary Outcome: AUC0-infinity (Area Under the Concentration-time Curve of BI 691751 in Plasma and Whole Blood Over the Time Interval From 0 Extrapolated to Infinity)
Description: AUC0-infinity (area under the concentration-time curve of BI 691751 in plasma and whole blood over the time interval from 0 extrapolated to infinity).
Time Frame: from day 1 to 31 days postdose relative to BI 691751 administration time: -2:00, 0:10, 0:20, 0:40, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00, 34:00, 47:00, 71:00, 95:00, 119:00, 143:00, 215:00, 287:00, 383:00, 551:00, 719:00h.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 691751 | IT + BI 691751
Number analyzed (Participants) | 20 | 20
nmol*h/L
  in plasma | 3160 (34.8) | 2360 (43.3)
  in whole blood | 27700 (29.6) | 24600 (29.6)
Statistical Analysis 1: Comparison: BI 691751 vs IT + BI 691751; gMean ratio of IT+BI 691751 to BI 691751 treatment (in plasma); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean ratio = 74.86, 90% CI 2-sided [62.946 to 89.035], Standard Error of Mean 32.4 — ratio of IT+BI 691751 to BI 691751 treatment. The standard error of the mean actually is the geometric coefficient of variance
Statistical Analysis 2: Comparison: BI 691751 vs IT + BI 691751; gMean ratio of IT+BI 691751 to BI 691751 treatment (in whole blood); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; gMean ratio = 88.19, 90% CI 2-sided [78.60 to 98.95], Standard Error of Mean 20.7 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From the 1st trial drug administration of a treatment until the 1st trial drug intake in the next treatment or until 31 days after the last administration of BI were assigned to the respective on-treatment phases (BI alone, loading IT, BI + further IT)
Description: More specifically, for: BI 691751 - up to 50 days, Loading IT - 3 days, BI + further IT - up to 47 days
Groups:
- BI 691751: 10 mg single dose oral administration with 240 mL water after intake of a standard meal. (only in the reference treatment period)
- Loading Itraconazole (IT): 200 mg of itraconazole (introductory treatment with itraconazole over three days, prior to the first administration of BI 691751 only in the test treatment period).
- BI 691751 + Further IT: 10 mg of BI 691751 in combination with multiple oral doses of itraconazole (only in the test treatment period after the introductory treatment with itraconazole alone over three days).
- Total BI 691751: total subjects with BI 691751 treatment (either BI 691751 alone or IT+BI 691751)
- Total on Treatment: combination of BI 691751, loading IT and BI 691751+ further IT.
Arm/Group | BI 691751 | Loading Itraconazole (IT) | BI 691751 + Further IT | Total BI 691751 | Total on Treatment
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes